CLINICAL TRIAL: NCT01147926
Title: A 12-week, Randomised, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy, Quality of Life, Safety and Tolerability of Prucalopride in Male Subjects With Chronic Constipation
Brief Title: Evaluation of Prucalopride in Male Subjects With Chronic Constipation.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD555-302; M0001-C302 (Other: Movetis); 2009-015719-42 (EudraCT Number)
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Male Subjects With Chronic Constipation
Keywords: Constipation; Male
MeSH Terms: conditions — Constipation | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Prucalopride (Active Comparator): 1 milligram (mg) or 2 mg
  Interventions: Drug: Prucalopride

INTERVENTIONS:
Drug: Placebo — Placebo matched to Prucalopride tablet orally once daily.
  Arms: Placebo
Drug: Prucalopride — Prucalopride 2 mg tablet orally once daily for subjects greater than or equal to (≥) 18 to less than (<) 65 years; 1 mg once daily orally for subjects ≥65 years, and in case of insufficient response, increased to 2 mg once daily orally at Week 2 or Week 4.
  Arms: Prucalopride

SUMMARY:
This is a multi-centre, randomised, parallel-group, double-blind, placebo-controlled phase III trial to evaluate the efficacy of prucalopride versus placebo over 12 weeks of treatment in male subjects with chronic constipation.

Furthermore the safety, tolerability, effect on quality of life and effect on symptoms of prucalopride will be assessed.

DETAILED DESCRIPTION:
In this phase III trial subjects will be screened and enter a 2-week run-in period (or a 3-week run-in period if the subject is using agents that influence bowel habit) during which the presence of constipation will be confirmed [the subject will complete an electronic daily diary (e-diary)]. At the start of run-in, all existing laxative medication will be withdrawn and subjects will be instructed not to change their diet or lifestyle during the trial. Subjects will be allowed to take a laxative [Dulcolax (bisacodyl)] as rescue medication during the trial, but only if they have not had a bowel movement (BM) for 3 or more consecutive days. An enema can only be used after unsuccessful use of Dulcolax (bisacodyl). No Dulcolax (bisacodyl) should be taken or enemas used between 48 hours before and 48 hours after the first intake of study medication.

After the run-in subjects will be randomly assigned to placebo or prucalopride in an equal ratio (1:1) if the subject fulfils the constipation criteria for inclusion. Randomisation will be stratified by country and by the average number of complete bowel movements (CBM) during run-in: 0 CBM/week and > 0 CBM/week.

Adult subjects (i.e. subjects ≥18 to <65 years of age) will take 2 mg prucalopride or matching placebo once daily before breakfast during the entire 12-week treatment period. Elderly subjects (i.e. subjects ≥65 years of age) will start at a dose of 1 mg prucalopride or matching placebo once daily before breakfast. In case of insufficient response, defined as an average of <3 spontaneous complete bowel movements (SCBM)/week during the preceding 2 weeks of treatment (i.e. since the previous visit) at Week 2 or Week 4, the daily dose has to be increased to 2 mg (or matching placebo). Once the dose is increased to 2 mg once daily the subject will stay on this dose for the remainder of the trial. After Week 4 (Visit 4) no changes in dose are allowed anymore.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male out-patient ≥18 years of age (no upper age limit).
2. Subject has a history of constipation. The subject reports an average of ≤ 2 SBM/week that result in a feeling of complete evacuation (SCBM) and one or more of the following for at least 6 months before the selection visit:

   1. Very hard (little balls) and/or hard stools for at least a quarter of the stools;
   2. Sensation of incomplete evacuation following for at least a quarter of the stools;
   3. Straining at defecation for at least a quarter of the time. This includes subjects who never have SBMs. The above criteria are only applicable for SBMs, i.e. BMs not preceded within a period of 24 hours by the intake of a laxative agent or by the use of an enema.
3. Subject agrees to stop his current laxative treatment and is willing to use rescue medication according to the rescue rule [Dulcolax® (bisacodyl)/enemas]
4. Subject's constipation is chronic.
5. Subject is able and willing to complete the questionnaires (if a validated version in the language of the subject is available) and the e-diary.
6. Subject voluntarily signs the written Informed Consent Form (ICF) in accordance with the regional laws/regulations, prior to the first trial-related activity.
7. Subject is willing to adhere to all trial requirements (amongst others colonoscopy/sigmoidoscopy, if required).

Exclusion Criteria:

1. Subjects in whom constipation is thought to be drug-induced.
2. Subjects using any disallowed medication
3. Subjects suffering from secondary causes of chronic constipation, such as:

   Endocrine disorders, e.g. hypopituitarism, hypothyroidism, hypercalcaemia, pseudohypoparathyroidism, pheochromocytoma or glucagon-producing tumours, unless these are controlled by appropriate medical therapy. Subjects with insulin-dependent diabetes mellitus should always be excluded, also if the subjects are under appropriate medical therapy; Metabolic disorders (e.g. porphyria, uraemia, hypokalaemia or amyloid neuropathy, unless these are controlled by appropriate medical therapy); Neurological disorders (e.g. Parkinson's disease, cerebral tumours, cerebrovascular accidents, multiple sclerosis, meningocele, aganglionosis, hypoganglionosis, hyperganglionosis, autonomic neuropathy or neuropathy due to chemotherapy, spinal cord injury, Chaga's disease, major depression); Surgery. Subjects with insulin-dependent diabetes mellitus should always be excluded, irrespective of whether the constipation started prior to or after the onset of diabetes.
4. Subjects with a significant history of cancer (i.e. less than a 5-year disease-free survival).
5. Subjects with intestinal perforation or obstruction due to structural or functional disorder of the gut wall, obstructive ileus, severe inflammatory conditions of the intestinal tract, such as Crohn's disease, and ulcerative colitis and toxic megacolon/megarectum. Results of an endoscopy or radiologic bowel evaluation is required to rule out polyps, cancer, stricture or other structural or organic disease:

   1. For patients ≤ 50 years: a flexible sigmoidoscopy or colonoscopy after the onset of constipation symptoms and within the previous 5 years;
   2. For patients > 50 years: a flexible sigmoidoscopy /double contrast barium enema or colonoscopy after the onset of constipation symptoms and within the previous 5 years.
   3. For subjects, regardless of age, even if results of this test are available within the previous 5 years but if the patient has alarm symptoms such as anemia, weight loss, heme positive stool, or rectal bleeding: a flexible sigmoidoscopy and double contrast barium enema or colonoscopy is needed after the onset of symptoms.
   4. If abnormalities have been detected during the sigmoidoscopy or colonoscopy e.g., because of polyps, the subject can be included in the trial if the polyps were removed. If clinically indicated, a repeat colonoscopy/sigmoidoscopy needs to be performed at latest within one week after the screening visit. If no barium enema with flexible sigmoidoscopy or a colonoscopic examination has been performed within the period as described above, the assessment is to be scheduled on the screening visit or within the week following screening. When it is clinically indicated that a repeat colonoscopy/sigmoidoscopy is needed to confirm results of a colonoscopy/sigmoidoscopy performed after the screening visit, the subject should be a screen failure.
6. Subjects with known serious illness: clinically significant cardiac, vascular, liver, pulmonary, or psychiatric disorders (as evaluated by the Investigator).
7. Subjects with any condition that in the opinion of the Investigator would complicate or compromise the trial or the well-being of the subject or evidence of clinically relevant pathology that could interfere with the trial results or put the subject's safety at risk.
8. Subjects known to have human immunodeficiency virus (HIV) infection or AIDS, hepatitis B or hepatitis C.
9. Subjects with impaired renal function, i.e. serum creatinine concentration >180 μmol/l or calculated creatinine clearance ≤30 ml/min, including subjects requiring dialysis.
10. Subjects with clinically significant abnormalities of haematology, urinalysis, or blood chemistry as determined by the Investigator. If the results of the haematology, biochemistry or urinalysis tests are not within the laboratory's reference ranges, the subject can be included only on the condition that the Investigator judges that the deviations are not clinically significant. This should be clearly recorded in the electronic Case Report Form (e-CRF).
11. Subjects with a known history of alcohol or drug abuse in the previous 6 months.
12. Subjects with lactose intolerance for whom it is expected that low doses of lactose can lead to diarrhoea, or a known allergy to ingredients or excipients of the trial medication.
13. Subjects who received an investigational drug in the 30 days preceding the run-in period of the trial.
14. Subjects who previously used prucalopride.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2010-09-23 (Actual); Primary Completion 2013-10-25 (Actual); Study Completion 2013-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (73):
- Belgium (6):
  - Gastro-Kliniek cvba, Antwerp
  - Cliniques Universitaires St Luc, Brussels
  - GP / Huisartsenpraktijk De Regenboog, Deurne
  - UZ Leuven Gasthuisberg, Leuven
  - CHU Sart Tilman, Liège
  - Private Practice, Wetteren
- 4 MHAT, Sofia, Bulgaria
- Czechia (9):
  - CCBR Czech Republic Brno, Brno
  - KKN a.s., Karlovy Vary
  - CCBR Czech Republic Pardubice, Pardubice
  - Universtiy Hospital Kralovske Vinhorady, Prague
  - MONSE s.r.o., Prague
  - Hospital Slany, Slaný
  - Orlickoustecka nemocnice, Ústí nad Orlicí
  - Krajska Nemocnice T. Bati a.s., Interni oddeleni - klinika IPVZ; Nemocnicni Lekarna, Zlín
  - Krajska Nemocnice T. Bati a.s., Zlín
- Denmark (3):
  - CCBR DK Aalborg, Aalborg
  - CCBR DK Ballerup, Ballerup Municipality
  - CCBR DK Vejle, Vejle
- France (13):
  - CHU - Hopital Nord, service gastro-enterologie et hepatologie, Amiens
  - ARK Clinical Research (Jean XXIII), Angers
  - ARK Clinical Research (Proust), Angers
  - ARK Clinical Research - Chanzy, Angers
  - ARK Clinical Research, Avrillé
  - Hopital Avicenne, Centre d'exploitation fonctionnelle et reducation digestive, Bobigny
  - Service de Gastroenterologie & INSERM CIC-P 803 - CHU de Dijon, Dijon
  - ARK Clinical Research, Le Plessis-Grammoire
  - Hôpital Edouard Herriot, Lyon
  - Hopital Archet 2- service gastro-enterologie et hepatologie, Nice
  - Hôpital Pontchaillou - Service des Maladies de l'Appareil Digestif, Rennes
  - Cabinet Médical, Thouars
  - ARK Clinical Research, Vendôme
- Germany (3):
  - emovis GmbH, Berlin
  - Gastroenterologie und Hepatologie am Johannisplatz, Leipzig
  - Fachartzpraxis für Innere Medizin, Wiesbaden
- Netherlands (7):
  - Meander Medisch Centrum, Amersfoort
  - VU Medisch Centrum, Amsterdam
  - PT&R / PreCare Trial & Recruitment, Beek
  - Ziekenhuis Gelderse Vallei, Ede
  - Maastricht Universitair medisch Centrum, Maastricht
  - Erasmus MC, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
- Poland (7):
  - Gabinet Lekarski Janusz Rudziński, Bydgoszcz
  - Instytut Medycyny Wsi im. Witolda Chodźki - Zaklad Endoskopowych Badań Kliniczncyh, Lublin
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Endoskopia Sp. z o.o., Sopot
  - Indywidualna Specjalistyczna Praktyka Lekarska w Dziedzinie Chirurgii Ogólnej i Gastroenterologii, Torun
  - Przychodnia Polskiej Fundacji Gastroenterologii Filia Nr 1 NZOZ, Warsaw
  - NZOZ Vivamed, Warsaw
- Romania (16):
  - CMI Dr. Lenghel Augustin, Oradea, Bihor County
  - Centrul Medical Valahia SRL, Ploieşti, Prahova
  - Spitalul Universitar de Urgenta Militar Central "Dr. Carol Davila", Bucharest, Sector 1
  - SC Quantum Medical Center SRL, Bucharest, Sector 1
  - Endocenter Medicina Integrativa SRL, Bucharest, Sector 2
  - SC Mediclass Sananova SRL, Bucharest, Sector 5
  - SC Cabinet Medical Dr. Blaj Stefan SRL, Bucharest, Sector 5
  - Centrul Medical Humanitas, Bucharest, Sector 6
  - Centrul Medical Tuculanu SRL, Timișoara, Timiș County
  - Centrul Medical Sana, Bucharest
  - Spitalul Clinic Judetean Cluj,Clinica Medicala I, Cluj-Napoca
  - Gastromedica SRL, Iași
  - Cabinet Medical Dr. Lokos Barna-Csaba, Miercurea-Ciuc
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
  - CMI de Gastroenterologie Dobru Daniela, Târgu Mureş
  - Policlinic Algomed SRL, Timișoara
- United Kingdom (8):
  - Oldfield Surgery, Bath
  - Avondale Surgery, Chesterfield
  - University Hospital & Warwickshire -, Coventry
  - County Durham & Darlington NHS Foundation Trust, Durham
  - Burbage Surgery, Hinckley
  - Townhead Research, Irvine
  - Wythenshawe Hospital, Manchester
  - Sherbourne Medical Centre, Royal Leamington Spa

REFERENCES:
- [Derived] Lembo A, Staller K, Boules M, Feuerstadt P, Spalding W, Gabriel A, Youssef A, Xie Y, Terreri B, Cash BD. Efficacy and safety of prucalopride in patients with chronic idiopathic constipation stratified by age, body mass index, and renal function: a post hoc analysis of phase III and IV, randomized, placebo-controlled clinical studies. Therap Adv Gastroenterol. 2024 Dec 10;17:17562848241299731. doi: 10.1177/17562848241299731. eCollection 2024. PMID 39664231
- [Derived] Staller K, Hinson J, Kerstens R, Spalding W, Lembo A. Efficacy of Prucalopride for Chronic Idiopathic Constipation: An Analysis of Participants With Moderate to Very Severe Abdominal Bloating. Am J Gastroenterol. 2022 Jan 1;117(1):184-188. doi: 10.14309/ajg.0000000000001521. PMID 34585675
- [Derived] Yiannakou Y, Piessevaux H, Bouchoucha M, Schiefke I, Filip R, Gabalec L, Dina I, Stephenson D, Kerstens R, Etherson K, Levine A. A randomized, double-blind, placebo-controlled, phase 3 trial to evaluate the efficacy, safety, and tolerability of prucalopride in men with chronic constipation. Am J Gastroenterol. 2015 May;110(5):741-8. doi: 10.1038/ajg.2015.115. Epub 2015 Apr 14. PMID 25869393

RESULTS

PARTICIPANT FLOW:
Groups:
- PRUCALOPRIDE: Prucalopride 2 milligram (mg) tablet orally once daily for subjects greater than or equal to (≥) 18 to less than (<) 65 years; 1 mg once daily orally for subjects ≥65 years, and in case of insufficient response, increased to 2 mg once daily orally at Week 2 or Week 4.
Period: Overall Study
Arm/Group | PLACEBO | PRUCALOPRIDE
Started | 187 | 187
Completed | 160 | 158
Not Completed | 27 | 29
Not completed — Subject Withdrew Consent | 9 | 10
Not completed — Adverse Event | 7 | 6
Not completed — Subject Non-Compliant | 5 | 4
Not completed — Principal investigator left hospital | 1 | 3
Not completed — Selection criteria not met | 3 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Sponsor's Decision | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Too busy, no time for study | 1 | 0
Not completed — Went on holiday | 0 | 1
Not completed — Colonoscopy result | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population included all subjects randomized into the study and who took at least 1 dose of investigational product (n = 370).
Groups:
- PRUCALOPRIDE: Prucalopride 2 mg tablet orally once daily for subjects ≥18 to <65 years; 1 mg once daily orally for subjects ≥65 years, and in case of insufficient response, increased to 2 mg once daily orally at Week 2 or Week 4.
- Total: Total of all reporting groups
Arm/Group | PLACEBO | PRUCALOPRIDE | Total
Number analyzed (Participants) | 186 | 184 | 370
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (16.28) | 58.4 (17.57) | 58.5 (16.91)
Age, Customized [Count of Participants; unit: Participants]
  Less than 65 years | 115 | 104 | 219
  Between 65 and 75 years | 39 | 43 | 82
  75 years and above | 32 | 37 | 69
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 186 | 184 | 370
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 10 | 10 | 20
  BULGARIA | 9 | 9 | 18
  CZECH REPUBLIC | 15 | 14 | 29
  DENMARK | 21 | 19 | 40
  FRANCE | 20 | 21 | 41
  GERMANY | 11 | 10 | 21
  NETHERLANDS | 5 | 5 | 10
  POLAND | 28 | 26 | 54
  ROMANIA | 57 | 56 | 113
  UNITED KINGDOM | 10 | 14 | 24

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects With an Average of ≥3 Spontaneous Complete Bowel Movements (SCBM) Per Week
Description: Spontaneous Bowel Movements defined as a bowel movement that is not preceded within a period of 24 hours by the intake of a laxative agent or by the use of an enema.
Time Frame: Over 12 week treatment period
Population: Modified Intent-to-treat Population (mITT) included all subjects randomized into the study except those excluded due to a major good clinical practice (GCP) breach at one site, who took at least 1 dose of the investigational product.
Measure: Number; unit: percentage of subjects
Arm/Group | PLACEBO | PRUCALOPRIDE
Number analyzed (Participants) | 181 | 177
percentage of subjects | 17.7 | 37.9
Statistical Analysis 1: Comparison: PLACEBO vs PRUCALOPRIDE; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Subjects With an Average Weekly Frequency of at Least 3 SCBM Per Week and an Increase of ≥ 1 SCBM Per Week for ≥ 75% of the 12-week Treatment Period and ≥ 75% of the Last Third of the 12-week Treatment Period
Time Frame: Over 12 week treatment period
Population: mITT
Measure: Number; unit: percentage of subjects
Arm/Group | PLACEBO | PRUCALOPRIDE
Number analyzed (Participants) | 181 | 177
percentage of subjects | 12.2 | 27.7

3. Secondary Outcome: Percentage of Subjects With an Increase of at Least 1 SCBM Per Week
Time Frame: Over 12 week treatment period
Population: mITT
Measure: Number; unit: percentage of subjects
Arm/Group | PLACEBO | PRUCALOPRIDE
Number analyzed (Participants) | 181 | 177
percentage of subjects | 45.3 | 53.7

4. Secondary Outcome: SCBM Per Week
Time Frame: Over 12 week treatment period
Population: mITT. Not all subjects in the mITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: SCBM/week
Arm/Group | PLACEBO | PRUCALOPRIDE
Number analyzed (Participants) | 172 | 170
SCBM/week | 1.8 (1.91) | 2.6 (2.40)

5. Secondary Outcome: Percent SBM With a Consistency of Normal and Hard/Very Hard
Description: Consistency measured using the 7-point Bristol scale where 1-2 indicate constipation (=hard/very hard), 3-4 are ideal stools (=normal), and 5-7 tending toward diarrhea.
Time Frame: Over 12 week treatment period
Population: mITT. Not all subjects in the mITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: percentage of SBM
Arm/Group | PLACEBO | PRUCALOPRIDE
Number analyzed (Participants) | 167 | 170
percentage of SBM
  Normal consistency | 50.8 (30.21) | 47.5 (31.70)
  Hard/Very hard consistency | 31.9 (29.86) | 26.9 (28.27)

6. Secondary Outcome: Percent SCBM With No Straining and Severe/Very Severe Straining
Description: Straining was evaluated on a 5-point scale (0=none, 1=mild, 2=moderate, 3=severe, or 4=very severe)
Time Frame: Over 12 week treatment period
Population: mITT. Not all subjects in the mITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: percentage of SBM
Arm/Group | PLACEBO | PRUCALOPRIDE
Number analyzed (Participants) | 167 | 170
percentage of SBM
  No straining | 9.5 (16.23) | 9.7 (17.40)
  Severe/Very severe straining | 23.7 (27.62) | 20.6 (27.33)

7. Secondary Outcome: Percent SBM With Sensation of Complete Evacuation
Time Frame: Over 12 week treatment period
Population: mITT. Not all subjects in the mITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: percentage of SBM
Arm/Group | PLACEBO | PRUCALOPRIDE
Number analyzed (Participants) | 167 | 170
percentage of SBM | 43.2 (32.90) | 46.7 (34.19)

8. Secondary Outcome: Time to First SCBM After Investigational Product Intake on Day 1
Time Frame: Day 1
Population: mITT.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | PLACEBO | PRUCALOPRIDE
Number analyzed (Participants) | 181 | 177
hours | 218.9 [143.93 to 291.43] | 110.3 [70.8 to 172.77]

9. Secondary Outcome: Bisacodyl Tablets Taken Per Week
Time Frame: Over 12 week treatment period
Population: mITT. Not all subjects in the mITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: Tablets/week
Arm/Group | PLACEBO | PRUCALOPRIDE
Number analyzed (Participants) | 172 | 170
Tablets/week | 1.0 (1.76) | 0.6 (1.56)

10. Secondary Outcome: Days With Rescue Medication Taken Per Week
Time Frame: Over 12 week treatment period
Population: mITT. Not all subjects in the mITT population had data for this outcome.
Measure: Mean (Standard Deviation); unit: Days/week
Arm/Group | PLACEBO | PRUCALOPRIDE
Number analyzed (Participants) | 172 | 170
Days/week | 0.6 (0.94) | 0.3 (0.69)

11. Secondary Outcome: Percent of Subjects With an Improvement of ≥ 1 Point on the Patient Assessment of Constipation - Symptom (PAC-SYM) Questionnaire Total Score at Final On Treatment Assessment
Description: The PAC-SYM is a validated 12-item questionnaire for the evaluation of severity of symptoms of constipation in subjects with constipation. Items are rated on a 5-point Likert scale: 0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe. Total score ranges from 0 to 48. Lower scores indicate improvement in symptoms. A 1-point improvement in PAC-SYM total score was considered clinically meaningful.
Time Frame: Over 12 week treatment period
Population: mITT. Not all subjects in the mITT population had data for this outcome.
Measure: Number; unit: percentage of subjects
Arm/Group | PLACEBO | PRUCALOPRIDE
Number analyzed (Participants) | 171 | 169
percentage of subjects | 30.4 | 34.9

12. Secondary Outcome: Percent of Subjects With an Improvement of ≥ 1 Point on the Patient Assessment of Constipation - Quality of Life (PAC-QOL) Total Score at Final On Treatment Assessment
Description: The PAC-QOL is a validated 28-item questionnaire for the evaluation of quality of life in subjects with constipation. Items are rated on a 5-point Likert scale: 0=not at all/none of the time, 1=a little bit/a little bit of the time, 2=moderately/some of the time, 3=quite a bit/most of the time, 4=extremely/all of the time. Total score ranges from 0-112. Lower scores indicate improvement in symptoms. A 1-point improvement in PAC-QOL total score was considered clinically meaningful.
Time Frame: Over 12 week treatment period
Population: mITT. Not all subjects in the mITT population had data for this outcome.
Measure: Number; unit: percentage of subjects
Arm/Group | PLACEBO | PRUCALOPRIDE
Number analyzed (Participants) | 171 | 169
percentage of subjects | 32.7 | 40.2

13. Secondary Outcome: Percent of Subjects on the Subject Global Evaluation on Severity of Constipation Score Rating Constipation as Severe to Very Severe at Final On-Treatment Assessment
Description: Subject was asked to rate the severity of his constipation using a 5-point Likert scale: 0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe
Time Frame: Over 12 week treatment period
Population: mITT. Not all subjects in the mITT population had data for this outcome.
Measure: Number; unit: percentage of subjects
Arm/Group | PLACEBO | PRUCALOPRIDE
Number analyzed (Participants) | 171 | 169
percentage of subjects | 30.4 | 21.9

14. Secondary Outcome: Percent of Subjects on the Subject Global Evaluation on Efficacy of Treatment Score Rating Treatment as Quite a Bit to Extremely Effective at Final On-Treatment Assessment
Description: The subject was asked to rate his global evaluation of the efficacy of treatment using the following 5-point scale: 0=not at all effective 1=a little bit effective 2=moderately effective 3=quite a bit effective 4=extremely effective.
Time Frame: Over 12 week treatment period
Population: mITT. Not all subjects in the mITT population had data for this outcome.
Measure: Number; unit: percentage of subjects
Arm/Group | PLACEBO | PRUCALOPRIDE
Number analyzed (Participants) | 171 | 169
percentage of subjects | 30.4 | 46.7

ADVERSE EVENTS:
Groups:
- PRUCALOPRIDE: Prucalopride 2 mg tablet orally once daily for subjects ≥18 to less than <65 years; 1 mg once daily orally for subjects ≥65 years, and in case of insufficient response, increased to 2 mg once daily orally at Week 2 or Week 4.
Arm/Group | PLACEBO | PRUCALOPRIDE
Serious Adverse Events (participants affected / at risk) | 4/186 | 1/184
Other Adverse Events (participants affected / at risk) | 21/186 | 37/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=186) | PRUCALOPRIDE (N=184)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
GLOTTIS CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=186) | PRUCALOPRIDE (N=184)
ABDOMINAL PAIN (Gastrointestinal disorders) | 11 (12) | 8 (11)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 12 (16)
NAUSEA (Gastrointestinal disorders) | 4 (4) | 11 (12)
HEADACHE (Nervous system disorders) | 7 (8) | 17 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.